CLINICAL TRIAL: NCT06449833
Title: Effect of Henagliflozein on Hepatic Fat Content in Patients With Type 2 Diabetes Mellitus and Nonalcoholic Fatty Liver Disease: A Multicenter, Randomized, Controlled Clinical Trial
Brief Title: Effect of Henagliflozein on Hepatic Fat Content in Patients With T2DM and NAFLD
Acronym: HHTN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023LX0120_GY
Record Dates: First submitted 2024-04-15; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-02

CONDITIONS: Type2 Diabetes Mellitus; Nonalcoholic Fatty Liver Disease
Keywords: Type 2 Diabetes Mellitus; Nonalcoholic fatty liver disease; Hepatic Fat Content; Henagliflozein; liver function
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — Metformin; Jentadueto

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Patients whose blood glucose are regulated by10 mg of Henagliflozein and metformin.
  Interventions: Drug: Henagliflozein and Metformin
- placebo (Placebo Comparator): Patients whose blood glucose are regulated by5mg of Linagliptin and metformin.
  Interventions: Drug: Linagliptin and Metformin

INTERVENTIONS:
Drug: Henagliflozein and Metformin — The experimental group will be treated with 10mg Henagliflozein and Metformin.
  Arms: intervention
Drug: Linagliptin and Metformin — The control group will be treated with 5mg Linagliptin and Metformin.
  Arms: placebo

SUMMARY:
This study focuses on the effects of Henagliflozein on hepatic fat content in patients with type 2 diabetes mellitus (DM) and nonalcoholic fatty liver disease (NAFLD). Sponsored by Zhujiang Hospital of Southern Medical University, this study is a multi-center, randomized, controlled clinical trial, aiming at exploring the difference in the reduction of liver fat content in the subjects compared with the control group after 24 weeks of treatment. Subjects from different medical centers diagnosed with T2DM and NAFLD will be randomly assigned to the treatment or control group in a 1:1 ratio, and subsequently initiate the intervention period of 24 weeks. In this trial, patients will be treated with 10 mg of Henagliflozein + metformin and 5 mg of Linagliptin + metformin as control, and the dose of metformin will be customized at 500-1500mg according to their individual blood glucose level. The check-points are set at the 8th, 16th and 24th week of the follow-up after the treatment, and nutritionists are available to provide dietary and exercise guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with type 2 diabetes within 5 years (According to the diagnostic criteria of WHO Diabetes Classification 2019)
2. Patients who are aware of the purpose of the trail, willing to participate in the trial and sign informed consent forms, and comply with all requirements (including those during follow-up and evaluation investigations)
3. Well-controlled blood glucose through diet and exercise intervention, or stable treatment with 1 or 2 types of hypoglycemic drugs (metformin, sulfonylurea, glinide, α-glycosidase inhibitor ) for at least 8 weeks with a half or full recommended maximum tolerated dose in instructions.
4. HbA1c: 7.0%-8.5%
5. Patients diagnosed with non-alcoholic fatty liver disease (According to the diagnostic criteria of Guidelines for Diagnosis and Treatment of Non-alcoholic Fatty Liver Disease 2010)

Exclusion Criteria:

1. Patients with type 1 diabetes, gestational diabetes or other special types of diabetes;
2. Patients with any acute, chronic complication or risk that may cause greater adverse effects than benefits through the trial; or receiving other treatment currently that may affect subjects' compliance or the objectivity of the end point of this trial; (1)Patients with serious acute complications of diabetes in the past 6 months (Eg. diabetic ketoacidosis, hyperosmotic hyperglycemia coma); (2)Patients with unstable proliferative retinopathy or maculopathy,severe diabetic neuropathy, intermittent claudication or diabetic foot in the past 6 months; (3)Patients with serious liver dysfunction and chronic kidney disease or disease of other systems (Eg. Acute and chronic pancreatitis, liver cirrhosis, nephrotic syndrome ect. ); and those who do not meet the requirements after being evaluated by professionals; (4)Have a history of myocardial infarction, unstable angina pectoris, stroke or transient ischemic attack, or underwent coronary angioplasty, percutaneous coronary stenting or coronary artery bypass grafting 6 months before the screening; or screening for congestive heart failure (New York Heart Association NYHA grade III and IV), unstable or acute congestive heart failure, or persistent arrhythmias believed to be life-threatening within the first 6 months of the trail; (5)Have a history of hemorrhagic stroke or ischemic stroke in the past 6 months, and was evaluated by the researchers as not suitable to participate in this clinical trial; (6)Have a history of hypertension and was not effectively controlled before screening: systolic blood pressure (SBP) ≥ 160mmHg and / or diastolic blood pressure (DBP) ≥ 100mmHg;
3. Have a history of other endocrine system diseases which affect glucose and lipid metabolism or have an effect on the body weight, such as: multiple endocrine adenomatosis, acromegaly, Cushing syndrome, hyperthyroidism;
4. Have a history of malignant tumour within 5 years before screening, except for local basal cell carcinoma of the skin after treatment；
5. Have a history of severe infection, trauma or major surgery within 3 months;
6. Have a history of drug abuse with 5 years, including repeated use of dependence-producing drug unrelated to medical purposes, including addictive and habitual drugs leading to physical and psychic dependence;
7. Have a history of participating any intervention drug or instrumental clinical trial 3 months before screening;
8. Have a history of severe anemia or need regular blood transfusion treatment;
9. Have a history of any medication or treatment below:

(1)Using drugs that may cause weight change 90 days before screening, including diuretics, weight-loss drug etc.; (2)Using drugs that may affect blood glucose for >1 week within 12 weeks, such as oral/intravenous glucocorticoid, growth hormone, estrogen/progesterone, high-dose diuretics, antipsychotic drugs, etc., but low-dose diuretics for antihypertensive purposes (hydrochlorothiazide < 25mg/d, indapamide < 1.5 mg/d) are not included in this restriction; (3)Had bariatric sugery or planning to have bariatric surgery; 10.The laboratory results of patients meet the following standards:

1. AlanineAminotransferase(ALT)and/oraspartateaminotransferase(AST) higher than 5 times of the upper limit of the normal value.
2. Glomerular Filtration Rate (eGFR) estimated by CKD-EPI formula < 40mL/ (min·1.73m2); 11.Patients are currently pregnant, breastfeeding or planning a pregnancy; 12.Have a history of infectious diseases such as hepatitis B (HBs-Ag), hepatitis C (HCV-Ab), pulmonary tuberculosis or sexually transmitted active diseases such as HIV and syphilis; 13.Have a history of using anti-NASH drugs (vitamin E, ursodeoxycholic acid, s-Adenosylmethionine, betaine, silymarin, gemdibrozil, anti-TNF therapy, probiotics, ect.) within 3 months before random grouping; 14.Having structural and functional genitourinary abnormalities prone to cause genitourinary infection; 15.Patients with abnormal hematologic system or any diseases that may cause hemolysis or unstable erythrocyte; 16.Have a history of using immunomodulators, such as biological agents, cyclophosphamide, cyclosporine, etc.; 17.Patients with MRI incompatible metal or magnetic implant, device or materials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The difference of liver fat content (magnetic resonance imaging proton density fat fraction,MRI-PDFF)) between the subjects and the control group. | 24 weeks

SECONDARY OUTCOMES:
The changes of liver enzymes (ALT). | 24 weeks
The changes of liver enzymes (AST). | 24 weeks
The changes of liver enzymes(GGT). | 24 weeks
The changes of hepatic fibrosis indexes(glutathione reductase). | 24 weeks
The changes of hepatic fibrosis indexes(total bile acid). | 24 weeks
The changes of hepatic fibrosis indexes(fibronectin). | 24 weeks
The changes of hepatic fibrosis indexes(N-terminal brain of type I procollagen.). | 24 weeks
The changes of hepatic fibrosis indexes(hyaluronic acid). | 24 weeks
The changes of hepatic fibrosis indexes(laminin). | 24 weeks
The changes of hepatic fibrosis indexes(type IV collagen). | 24 weeks
The changes of hepatic fibrosis indexes(glycocholic acid.). | 24 weeks
Changes of visceral fat volume. | 24 weeks
Changes of subcutaneous fat volume. | 24 weeks
Changes of fasting blood glucose. | 24 weeks
Changes of fasting insulin. | 24 weeks
Changes of HbA1c. | 24 weeks
Changes of (HOMA-R). | 24 weeks
Blood lipid index(TC). | 24 weeks
Blood lipid index(TG). | 24 weeks
Blood lipid index(HDL-C). | 24 weeks
Blood lipid index(LDL-C). | 24 weeks
Changes of body weight. | 24 weeks
Changes of BMI. | 24 weeks
Changes of waist circumference. | 24 weeks
Changes of hip circumference. | 24 weeks
Changes of WHR. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hong Chen, MD, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China